CLINICAL TRIAL: NCT00659308
Title: Amniotic Membrane and Anterior Stromal Puncture: a Comparative Study in the Treatment of Symptomatic Bullous Keratopathy
Brief Title: Amniotic Membrane and Anterior Stromal Puncture to the Treatment of Symptomatic Bullous Keratopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Fabiana Paris, Federal University of Sao Paulo
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: cep0728/02
Record Dates: First submitted 2008-04-14; First posted 2008-04-16 (Estimated); Last update posted 2008-04-16 (Estimated); Status verified 2008-01

CONDITIONS: Bullous Keratopathy
Keywords: pain; bullous keratopathy; amniotic membrane; anterior stromal puncture
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: amniotic membrane transplantation — patients are submitted to amniotic membrane transplantation
Procedure: anterior stromal puncture — the other group is submitted to anterior stromal puncture

SUMMARY:
The purpose of this study is to determine whether amniotic membrane transplantation is as effective as anterior stromal puncture in the relief of symptomatic bullous keratopathy.

DETAILED DESCRIPTION:
Patients with symptomatic bullous keratopathy were randomized in 2 groups and submitted to amniotic membrane transplantation or anterior stromal puncture. The follow up was made with 1, 3, 6 and 12 months. Evaluation included complete ophthalmologic exam, esthesiometry, pachymetry, impression cytology and evaluation of pain.

ELIGIBILITY:
Inclusion Criteria:

* bullous keratopathy

Exclusion Criteria:

* age under 18 years old
* asymptomatic bullous keratopathy
* corneal infection
* ocular hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2005-06; Primary Completion 2005-07 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fabiana Paris, MD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Federal University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Pires RT, Tseng SC, Prabhasawat P, Puangsricharern V, Maskin SL, Kim JC, Tan DT. Amniotic membrane transplantation for symptomatic bullous keratopathy. Arch Ophthalmol. 1999 Oct;117(10):1291-7. doi: 10.1001/archopht.117.10.1291. PMID 10532436
- [Background] Gomes JA, Haraguchi DK, Zambrano DU, Izquierdo Junior L, Cunha MC, de Freitas D. Anterior stromal puncture in the treatment of bullous keratopathy: six-month follow-up. Cornea. 2001 Aug;20(6):570-2. doi: 10.1097/00003226-200108000-00003. PMID 11473154